CLINICAL TRIAL: NCT01640821
Title: Dissemination of the "Choisir de Maigrir?" Program in Health and Social Service Centers in Québec: Evaluation of Its Implementation and Impact on Lifestyle Habits and Well-being
Brief Title: Dissemination of the "Choisir de Maigrir?" Program
Acronym: CHOIX-CSSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Véronique Provencher, Professeur sous octroi, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-ASSS-MTL-10-001
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Obesity
Keywords: Health-At-Every-Size intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (CdM?) (Experimental): This group will be composed of women that are seeking help for weight-related problems that have been referred to the CdM? program.
  Interventions: Behavioral: CdM? program
- Control group (No Intervention): This group will be composed of women that are seeking help for weight-related problems but that are actually on the waiting list for participating to the CdM? program.

INTERVENTIONS:
Behavioral: CdM? program — The program is conducted in small groups of 12 to 15 women for 14 weekly sessions (13 3h-evening sessions and 1 intensive-day session of 6 hours). Two health professionals (a registered dietician and a social worker or psychologist) lead the group. Sessions include lectures, guided self-examination and observations, group discussions, and practical exercises. Different topics are discussed during sessions such as enjoyment of physical activity and healthy nutrition, setting realistic objectives with regard to weight loss, and acceptation of their own and others' body image. A weekly food diary and group discussions are used to facilitate the recognition of internal cues of hunger and satiety and the identification of external influences on eating behaviors and food intake.
  Arms: Intervention group (CdM?)

SUMMARY:
The Québec government launched in October 2006 an action plan (PAG) to reduce the prevalence of overweight and obesity among young people and adults by 2012. One of the five priorities of the PAG is to improve health services for individuals with weight-related issues. The development and implementation of sustainable weight-control strategies however remains a challenge, since weight loss is often regained by the majority of individuals over time. "Health-At-Every-Size" (HAES) interventions, which are mainly focusing on health rather that weight, have been proposed as an interesting alternative for individuals, mainly women, who are struggling with weight-related issues. Based on the HAES, "Choisir de maigrir?" (CdM?) program has been clearly identified by the PAG as one of the actions for improving health services and Quebec's government has already started a massive dissemination of the CdM? program in CSSS of Québec. In that context, it becomes imperative to rapidly assess the effectiveness and readiness of the program for a broad dissemination. The present research proposal falls directly within the scope of the PAG recommendation and the investigators general objective is to develop a population-based understanding of the effectiveness of the CdM? program in Quebec's CSSS by documenting the effects of the program on women's health in a natural setting.

DETAILED DESCRIPTION:
The impact of "CdM?" will be assessed with each CSSS at three time points: at baseline (T=1), at the end of the intervention period (T=2), and at 1-y post-intervention (T=3). While data collection instructions and assessment materials will be provided by the research team, administration of the CdM? program will be totally under the responsibility of each CSSS, so that the program will occur outside of the research team control. Validated questionnaires will be used to assess nutritional profile, physical activity level, and psychosocial variables among the participants (N=168). Weight, height and waist circumference will also be measured for each participant. In order to ensure that our results are not due to the effect of time, women on a waiting list for CdM? program, will be recruited (N=84) for the short-term effect. All these data will be treated using sophisticated analyses strategies.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years old and over
* Seeking help for weight-related problems

Exclusion Criteria:

* Considering the natural setting of the present study and the fact that the program is occurring outside of the applicants' control, no stringent exclusion criteria will be determined.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Food habits | Up to one year post-intervention
  To evaluate the impact of the CdM? program on food habits for all women will be conducted at three time points: at baseline (T=1), at the end of the intervention period (T=2), and at 1-y post-intervention (T=3).

SECONDARY OUTCOMES:
Eating behaviors | Up to one year post-intervention
  To evaluate the impact of the CdM? program on eating behaviors.
Physical activity | Up to one year post-intervention
  To evaluate the impact of the CdM? program on physical activity.
Well-being | Up to one year post-intervention
  To evaluate the impact of the CdM? program on well-being.
Weight | Up to one year post-intervention
  To evaluate the impact of the CdM? program on weight.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Provencher, Ph.D., Principal Investigator — Laval University
Locations (1):
- Institute of Nutraceuticals and Functionnal Foods (INAF), Québec, Quebec, Canada